CLINICAL TRIAL: NCT03038984
Title: Are Rates of Colectomies, Resections, Mortalities and Cancer Reduced by Home Monitoring of IBD Patients Tightly on Demand or Every 3 Months by Fecal Calprotectin and Disease Activity?
Brief Title: Are Rates of Colectomies, Resections, Mortalities and Cancer Reduced by Home Monitoring of IBD Patients ?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Dorit Vedel Ankersen, PhD student, Msc food science and Msc Clinical nutrition, Nordsjaellands Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-15005603
Record Dates: First submitted 2017-01-24; First posted 2017-02-01 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD; Telemedicine; At-home monitoring; Disease activity; fecal calprotectin; Total inflammation burden; 11 years follow up
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: 120 IBD patients has been randomized to screen for disease activity and FC either OD or every 3 months. 60 patients in each group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Every 3 months (Experimental): screening every 3rd month: (home monitoring: FC and DA)
  Interventions: Behavioral: At Home Screening procedure every 3 months
- On demand (Active Comparator): screening On demand: (home monitoring: FC and DA)
  Interventions: Behavioral: At Home Screening procedure On demand

INTERVENTIONS:
Behavioral: At Home Screening procedure On demand — Home monitoring is a supportive treatment. Patients are randomized to screen themselves on demand
  Arms: On demand
Behavioral: At Home Screening procedure every 3 months — Home monitoring is a supportive treatment. Patients are randomized to screen themselves every 3 months
  Arms: Every 3 months

SUMMARY:
This study is a side protocol/extension of 10 years of ClinicalTrials.gov ID: NCT02492555. The purpose of this study is to determine if the IBD patients doing home monitoring (screening themselves on demand (OD) or every 3 months) have relative reduced rates of colectomies, resections, mortalities and cancer after 11 years of web monitoring. The IBD patients are self-monitoring by web apps consisting of a short disease activity questionnaire (DA) and fecal calprotectin (FC) on any smart phone.

DETAILED DESCRIPTION:
This study is a side protocol/extension of 10 years of ClinicalTrials.gov ID: NCT02492555. Among 2.500 IBD patients the investigators have consecutively from the Gastroenterology out-patient clinic at North Zealand University Hospital recruited in total 120 in the study.

At the out-patient consultation IBD patients has been informed about the project and the IBD eHealth nurse has ensured that no exclusion criteria was met by the patients.

Inclusion criteria:

IBD patients in remission, SCCAI ≤ 2 (Simple Clinical Colitis Activity Index )) or HBI < 5 (Harvey & Bradshaw Activity Index ) or in mild to moderate disease activity ( SCCAI 3-4, HBI < 16) IBD patients who can read, speak and understand Danish. IBD patients that can take advantage of the Internet and wireless network. 18 years or older.

Exclusion criteria:

IBD patients with severe disease activity HB > 16 SCCAI ≥ 5 IBD patients with social, medical or psychological issues of a more complex character. IBD patients with particularly complex issues such as drug and alcohol problems, severe mental / psychiatric disorders and / or serious social impact.IBD patients who cannot attend due language barrier or cognitive disorder. Age less than 18.

When the patient has agreed to participate in the study, randomized to either OD or 3. Months (This has been done ClinicalTrials.gov ID: NCT02492555)

Patients log in to www.noh.constant-care.dk at least once every 3rd months throughout the project period of 11 years in total (2015-2026). When the patient log in to the telemedicine platform the following scorings must be filled out:

1. - Disease activity (DA), respectively SCCAI or HBI.
2. - Quality of life assessment, s-IBDQ
3. - FACIT (Fatigue score)
4. - MARS ( Medical Adherence Rating Scale)
5. - FC, fecal calprotectin mg / kg measured by the patient's own SMART phone, rapid home test.

If the patients prefer to send the fecal samples for test, it will be analyzed in the ehealth gastro lab. at the hospital with a SMART phone as well.

The results of the scoring systems will appear to the health care professionals and patients in a traffic light manner (red, yellow and green).

If the patient experiences a recurrence of the disease, it moves from green to either yellow or red area in the traffic graph, and patient will further be instructed to contact Gastro medical clinic project nurse for an early consultation and decision on further treatment initiative. This will also be indicated at the patient's website. If alarm symptoms occurs patients are instructed to contact the project nurse. Thus patients are treated in accordance to national and international guideline. By screening of the inflammation burden (web algorithm), the decision is moving forward.

Patients logging in on demand, indicate disease activity, quality of life and FC at the start, and subsequently when needed and at the end of the study (after 11 years from inclusion).

At relapse, disease activity score and FC is settled and repeated no later than 7 days here after. When the patient has reached remission (green) a new DA and FC test should be performed to verify the remission.

The purpose of this study is to determine if the IBD patients doing home monitoring have relative reduced rates of colectomies, resections, mortalities and cancer after 11 years of web monitoring. Relative reduced rates of colectomies etc. means - relative to standard care but also if there is a difference between the two web screening procedures on these endpoints.

ELIGIBILITY:
Inclusion Criteria:

* IBD patients in remission, SCCAI ≤ 2 (Simple Clinical Colitis Activity Index )) or HBI < 5 (Harvey & Bradshaw Activity Index ) or in mild to moderate disease activity ( SCCAI 3-4, HBI < 16). IBD patients who can read, speak and understand Danish. IBD patients that can take advantage of the Internet and wireless network.

Exclusion Criteria:

* IBD patients with severe disease activity HB > 16 SCCAI ≥ 5. IBD patients with social, medical or psychological issues of a more complex character. IBD patients with particularly complex issues such as drug and alcohol problems, severe mental / psychiatric disorders and / or serious social impact.IBD patients who cannot attend due language barrier or cognitive disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
colectomies | 11 years
  Number of colectomies
resections | 11 years
  Number of resections
mortalities | 11 years
  Number of deaths
cancer | 11 years
  cancer rates

SECONDARY OUTCOMES:
Hospitalizations | 11 years
  number of hospitalizations and days
FC (Fecal Calprotectin) area under the curve (AUC) | 11 years
  Both AUC total, but also as a red >600 mg/kg, yellow (200-600 mg/kg) and green (below 200mg/kg ) AUC will be performed from the individualized curves
Simple clinical colitis activity index (SCCAI): area under the curve (AUC) | 11 years
  Both AUC total, but also as a red >5, yellow (2-4) and green (< 2 ) AUC will be performed from the individualized curves
Harvey-Bradshaw index (HBI): area under the curve (AUC) | 11 years
  Both AUC total, but also as a red >16 , yellow (6-16) and green (≤5) AUC will be performed from the individualized curves
Disease course, Copenhagen IBD Disease course Type | 11 years
  Based on epidemiology four figures have been developed to describe disease-course of IBD. These figures have been used in a retrospective study (Maagaard et al. 2016) to measure change in Disease course.The four figures depicting different types of disease courses is described as follows:
  1. Mild IBD with indolent course
  2. Mild IBD with aggressive course
  3. Chronic IBD with continuous course
  4. Chronic IBD with intermittent course The patients have to choose one figure representing their disease course type the best at inclusion and 11 years later

CONTACTS AND LOCATIONS:
Overall Officials: Pia Munkholm, Professor, Study Director — North Zealand University Hospital

IPD SHARING:
Plan to Share IPD: No